CLINICAL TRIAL: NCT07393451
Title: A Randomized, Double-blind, Placebo, Parallel-Controlled, Multicenter Phase 2a Clinical Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of SIM0278 in Subjects With Active Lupus Nephritis
Brief Title: A Multicenter Phase 2a Clinical Study to Evaluate SIM0278 in Subjects With Active Lupus Nephritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0278-202
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Cohort 1- Test group
  Interventions: Drug: SIM0278 injection
- Control group (Experimental): Cohort 2- Control group
  Interventions: Drug: SIM0278 injection

INTERVENTIONS:
Drug: SIM0278 injection — Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled multicenter clinical study to evaluate the efficacy, safety, and pharmacokinetics of SIM0278 in adult (18-75 years) subjects with active LN suitable for systemic therapy.

Approximately 60 subjects with active LN are planned to be enrolled and randomized 1: 1 to SIM0278 or placebo.

The study consists of 3 phases: screening, double-blind treatment, and safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥ 40.0 kg
2. SLE was diagnosed according to 2019 American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) classification criteria.
3. Subjects must be receiving or willing to initiate induction therapy for LN. Induction therapy, defined as including high-dose glucocorticoids and MMF, should be initiated within 60 days or on the same day prior to baseline.

Exclusion Criteria:

1. Previous or current nephropathy (except LN) that, in the opinion of the investigator, may interfere with the LN assessment and interfere with the assessment of disease activity (e.g., diabetic nephropathy). The subject was unable or unwilling to provide written informed consent and/or to comply with study procedures.
2. Severe renal impairment: a) oliguria (defined as recorded urine volume < 400 mL/24 h), or b) end-stage renal disease (ESRD) requiring dialysis or transplantation.
3. Previous induction therapy for MMF/MPS was considered by the investigator to have failed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving an overall renal response (complete renal response (CRR) + partial renal response (PRR)) at Week 52 | At Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No